CLINICAL TRIAL: NCT02083705
Title: Chest Compression and Sustained Inflation for Asystole or Bradycardia in Newborn Infants
Brief Title: Chest Compression and Sustained Inflation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00034524_CC
Record Dates: First submitted 2014-01-13; First posted 2014-03-11 (Estimated); Results first posted 2024-09-20 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Newborn Infants Having Asystole or Bradycardia at Birth
Keywords: Chest compression, Delivery Room, NICU,
MeSH Terms: interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SI+CC (Experimental): Chest compression will be superimposed by sustained inflations during CPR:
  "CC+SI group" Infants randomized in the SI group requiring CC, would receive CC at a rate of 90/min during an SI with a duration of 20sec (CC+SI). After 20 sec the SI will be interrupted for 1 sec and the next SI will be started for another 20sec13. Throughout this time CC is continued until ROSC. Every 45 sec (approximately 2 SIs) the clinical team would assess for changes in heart rate. CC+SI was continued until ROSC.
  Interventions: Procedure: CC+SI
- 3:1 CPR (Active Comparator): CPR using 3:1 C:V ratio:
  "3:1 C:V group" Infants randomized into the "3:1 group" requiring CC, would received CC using the current 3:1 C:V ratio recommend in the neonatal resuscitation guidelines16. Every 45 sec the clinical team would assess heart rate. 3:1 C:V CPR was continued until ROSC.
  Interventions: Procedure: 3:1 CPR

INTERVENTIONS:
Procedure: CC+SI — Chest compression will be superimposed by sustained inflation during CPR
  Arms: SI+CC
Procedure: 3:1 CPR — CPR using 3:1 ratio (control group)
  Arms: 3:1 CPR

SUMMARY:
Guidelines on neonatal resuscitation recommend 90 chest compressions (CC) and 30 manual inflations (3:1) per minute in newborns. The study aimed to determine if CC s during sustained inflations (SI) improves recovery of asphyxiated newborns compared to coordinated 3:1 resuscitation.

ELIGIBILITY:
Inclusion Criteria:

Newborn infants with asystole Newborn infants with bradycardia

Exclusion Criteria:

-

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Schmolzer GM, O Reilly M, Fray C, van Os S, Cheung PY. Chest compression during sustained inflation versus 3:1 chest compression:ventilation ratio during neonatal cardiopulmonary resuscitation: a randomised feasibility trial. Arch Dis Child Fetal Neonatal Ed. 2018 Sep;103(5):F455-F460. doi: 10.1136/archdischild-2017-313037. Epub 2017 Oct 7. PMID 28988159

RESULTS

PARTICIPANT FLOW:
Groups:
- SI+CC: Chest compression will be superimposed by sustained inflations during CPR:
  "CC+SI group" Infants randomized in the SI group requiring CC, would receive CC at a rate of 90/min during an SI with a duration of 20sec (CC+SI). After 20 sec the SI will be interrupted for 1 sec and the next SI will be started for another 20sec13. Throughout this time CC is continued until ROSC. Every 45 sec (approximately 2 SIs) the clinical team would assess for changes in heart rate. CC+SI was continued until ROSC.
  CC+SI: Chest compression will be superimposed by sustained inflation during CPR
- 3:1 CPR: CPR using 3:1 C:V ratio:
  "3:1 C:V group" Infants randomized into the "3:1 group" requiring CC, would received CC using the current 3:1 C:V ratio recommend in the neonatal resuscitation guidelines16. Every 45 sec the clinical team would assess heart rate. 3:1 C:V CPR was continued until ROSC.
  3:1 CPR: CPR using 3:1 ratio (control group)
Period: Overall Study
Arm/Group | SI+CC | 3:1 CPR
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SI+CC | 3:1 CPR | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 4 | 9
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Time Needed to Achieve Return of Spontaneous Circulation
Description: We aim to reduce time needed to achieve Return of Spontaneous Circulation. This should be achieved by the experimental chest compression technique
Time Frame: within the first 10 minutes after birth
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | SI+CC | 3:1 CPR
Number analyzed (Participants) | 5 | 4
seconds | 31 (9) | 138 (72)
Statistical Analysis 1: Comparison: SI+CC vs 3:1 CPR; We hypothesised that during neonatal CPR, CC+SI will reduce the time needed to achieve ROSC. Our aim was to examine if CC+SI reduces ROSC compared with 3:1 C:V CPR in preterm infants <33 weeks of gestation. For this pilot study, based on the local incidence of CPR in preterm neonates, a convenient sample size of five patients per group was enrolled. Our primary outcome was time to achieve ROSC measured using ECG; Test type: Superiority; p = 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: within 6 months
Arm/Group | SI+CC | 3:1 CPR
All-Cause Mortality (participants affected / at risk) | 2/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 4/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SI+CC (N=5) | 3:1 CPR (N=4)
Air leak (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Intraventricular haemorrhage all grades (Nervous system disorders) | 1 (1) | 4 (4)
Intraventricular haemorrhage grade >3 (Nervous system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes